CLINICAL TRIAL: NCT00643695
Title: Efficacy of an Exercise Intervention to Decrease Depressive Symptoms in Veterans With Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patricia Taylor-Young, Nurse Scientist, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02101
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C; Depression
Keywords: hepatitis C; depression; exercise
MeSH Terms: conditions — Hepatitis C; Depression; Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Home-based walking program
  Interventions: Behavioral: Home-based walking program
- 2 (Other): educational intervention
  Interventions: Other: Educational intervention

INTERVENTIONS:
Behavioral: Home-based walking program — The exercise intervention is a 12 week home-based exercise program. Ideally Individuals will walk for 30 minutes, at a moderate intensity, a minimum of three times per week. However, the duration and relative intensity will be tailored for each individual.
  Arms: 1
Other: Educational intervention — Participants in the control group will receive a packet of information regarding hepatitis C
  Arms: 2

SUMMARY:
In this study, depressed veterans with hepatitis C will be randomly assigned to the control group or to the exercise intervention group. The exercise intervention is designed to begin slowly for most participants and to progress within each participant's target heart rate range for moderate intensity exercise. The exercise intervention is a 12 week home based walking program. Ideally individuals will walk for 30 minutes, at a moderate intensity, a minimum of three times per week. However, the duration and relative intensity will be tailored for each individual.

Central Hypothesis Veterans who receive the exercise intervention will be significantly less symptomatic for depression than veterans in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 or older
* Documentation of positive hepatitis C status as indicated by a detectable HCV viral load by polymerase chain reaction
* Mild to moderate depressive symptoms as evidenced by a BDI II score of ≥ 14
* Able to read and understand English
* Written/signed informed consent specific to this protocol
* Being sedentary that is , less than 30 minutes of planned low to moderate intensity exercise 2 days per week

Exclusion Criteria:

* Suicidal ideations
* Current interferon therapy or planning to begin interferon therapy during the next three months
* Diagnosis of Bipolar disorder, Schizophrenia, or Post Traumatic Stress Disorder
* Any medical condition, disorder, or medication that contraindicates participation in a mild to moderate intensity walking program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Reduction of symptoms of depression as measured by the Beck Depression Inventory II (BDI-II) | 12 weeks

SECONDARY OUTCOMES:
Reduction in symptoms of fatigue as measured by the Brief Fatigue Inventory (BFI) | 12 weeks
reduce the reported level of chronic pain | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Taylor-Young, PhD, RN,FNP, Principal Investigator — Portland VA Medical Center
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States